CLINICAL TRIAL: NCT01424696
Title: Baby Observational and Nutritional Study (BONUS)
Brief Title: Baby Observational and Nutritional Study
Acronym: BONUS
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Bonnie Ramsey, Professor, Seattle Children's Hospital
Other Study IDs: BONUS-IP-11; R01DK095738 (NIH)
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Cystic Fibrosis; Growth Failure; Exocrine Pancreatic Insufficiency
Keywords: growth measures; nutritional status; pulmonary infection; inflammatory markers; pancreatic enzyme replacement therapy
MeSH Terms: conditions — Cystic Fibrosis; Failure to Thrive; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * serum and/or plasma
  * urine
  * stool
  * oropharyngeal swab (OP swab)
  * saliva
  * sweat
  * buccal brushings
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cystic Fibrosis in 1st 3 months of life: Early Diagnosis: Children diagnosed with CF in first 3 months of life

SUMMARY:
Cystic fibrosis (CF) is a life-shortening disease that causes breathing and digestive problems, but can now be diagnosed at the time of birth. Lung function is very hard to measure in infants, but growth is not. In this study the investigators aim to define growth in infants with CF in the first year of life with research quality precision and to understand factors that interfere with good growth.

Pancreatic enzyme replacement therapy (PERT) will be also be studied in a subgroup of infants. Two different doses of PERT will be evaluated for improving fat and nitrogen absorption in infants with CF.

DETAILED DESCRIPTION:
Newborn screening (NBS) for cystic fibrosis (CF) has decreased the prevalence of malnutrition in infancy, but suboptimal nutrition still persists. In one study, 60% of infants diagnosed by NBS achieved their birth weight percentile by two years of age, while 40% did not. The many factors that contribute to this poor growth have not been defined and persist despite pancreatic enzyme supplementation. Although published guidelines for the clinical management of infants with cystic fibrosis in the U.S. and Europe exist, there is an alarming scarcity of evidence to dictate care. In order to proceed with large scale randomized studies to evaluate the range of interventions for infants with CF, we need to not only develop precise techniques for measuring growth but also pursue unexplored factors that may contribute to poor growth.

This is a multi-center observational clinical study with a nested interventional PERT sub-study. The observational study was designed to follow in a prospective manner incident cases of CF for up to 12 months. The PERT sub-study is a randomized, double-blind, crossover sub-study designed to evaluate the efficacy and safety of two doses of PERT (pancreatic enzyme replacement therapy) for improving coefficient of fat absorption (CFA) in the stool of infants with CF. The PERT sub-study was unable to enroll and closed. No results available.

ELIGIBILITY:
Observational Study

Inclusion Criteria:

1. Signed informed consent
2. Males or females no more than three and one half (3.5) months of age at enrollment
3. Documentation of a CF diagnosis as evidenced by:

   1. One or more of the following: one or more clinical features consistent with the CF phenotype OR a positive newborn screening (NBS) OR a positive pre-natal screen

      AND
   2. One or more of the following: sweat chloride ≥ 60 mEq/liter by quantitative pilocarpine iontophoresis test (QPIT) OR two well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
4. Enrolled in the Cystic Fibrosis Foundation Patient Registry. (Patients may enroll in the Registry at Enrollment Visit if not previously enrolled.)

Exclusion Criteria:

1. Children unable to take full oral feeds
2. Any serious or active medical condition, which in the opinion of the investigator, contributes to malabsorption, interferes with normal growth, or would otherwise interfere with subject's treatment, assessment, or compliance with the protocol.
3. Gestational age less than 35 weeks and/or birth weight < 2.5 kg.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants diagnosed with CF who attend regular clinic visits during the first year of life
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2011-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incremental gain in weight, length, and head circumference | one year
  To define and describe incremental weight gain and linear growth in the first year of life utilizing research quality growth measures that will be applicable as efficacy outcomes for future interventional studies in infants with CF

CONTACTS AND LOCATIONS:
Overall Officials: Drucy Borowitz, MD, Principal Investigator — State University of New York at Buffalo; Daniel Leung, MD, Principal Investigator — Baylor College of Medicine; James Heubi, MD, Principal Investigator — University of Cincinnati; Daniel Gelfond, MD, Principal Investigator — Women & Children's Hospital of Buffalo
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Colorado, Aurora, Colorado
  - Emory CF Center, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Iowa City University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital CF Care Center, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - State University of New York at Buffalo, Buffalo, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt CF Center, Nashville, Tennessee
  - Austin Children's Chest Associates, Austin, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Sathe M, Huang R, Heltshe S, Eng A, Borenstein E, Miller SI, Hoffman L, Gelfond D, Leung DH, Borowitz D, Ramsey B, Freeman AJ. Gastrointestinal Factors Associated With Hospitalization in Infants With Cystic Fibrosis: Results From the Baby Observational and Nutrition Study. J Pediatr Gastroenterol Nutr. 2021 Sep 1;73(3):395-402. doi: 10.1097/MPG.0000000000003173. PMID 34016873
- [Derived] Goetz D, Kopp BT, Salvator A, Moore-Clingenpeel M, McCoy K, Leung DH, Kloster M, Ramsey BR, Heltshe SH, Borowitz D. Pulmonary findings in infants with cystic fibrosis during the first year of life: Results from the Baby Observational and Nutrition Study (BONUS) cohort study. Pediatr Pulmonol. 2019 May;54(5):581-586. doi: 10.1002/ppul.24261. Epub 2019 Jan 22. PMID 30672141
- [Derived] LeGrys VA, Moon TC, Laux J, Accurso F, Martiniano SA. A multicenter evaluation of sweat chloride concentration and variation in infants with cystic fibrosis. J Cyst Fibros. 2019 Mar;18(2):190-193. doi: 10.1016/j.jcf.2018.12.006. Epub 2018 Dec 21. PMID 30583934
- [Derived] Kopp BT, Joseloff E, Goetz D, Ingram B, Heltshe SL, Leung DH, Ramsey BW, McCoy K, Borowitz D. Urinary metabolomics reveals unique metabolic signatures in infants with cystic fibrosis. J Cyst Fibros. 2019 Jul;18(4):507-515. doi: 10.1016/j.jcf.2018.10.016. Epub 2018 Nov 23. PMID 30477895
- [Derived] Gelfond D, Heltshe SL, Skalland M, Heubi JE, Kloster M, Leung DH, Ramsey BW, Borowitz D; BONUS Study Investigators. Pancreatic Enzyme Replacement Therapy Use in Infants With Cystic Fibrosis Diagnosed by Newborn Screening. J Pediatr Gastroenterol Nutr. 2018 Apr;66(4):657-663. doi: 10.1097/MPG.0000000000001829. PMID 29176494